CLINICAL TRIAL: NCT01662115
Title: Does Nicotine Gum Enhance Bowel Recovery After Colorectal Surgery?
Brief Title: Nicotine Gum Recovery After Colorectal Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has been terminated due linability to recruit the targeted participants. Aimed for 300 participants and only 4 were enrolled after 1 year.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Weiss, DIO and Chairman of Graduate Medical Education at Cleveland Clinic Florida,, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CRS-2012-05
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Post-operative Ileus
Keywords: ILEUS
MeSH Terms: conditions — Ileus | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nicotine gum (Active Comparator): 100 subjects who will actually get the intervention medication
  Interventions: Drug: Nicotine gum
- regular chewing gum (Sham Comparator): 100 subjects who will be part of a control group
  Interventions: Other: Regular chewing gum
- No gum (No Intervention): 100 subjects who will not get neither the intervention nor the placebo gum.

INTERVENTIONS:
Drug: Nicotine gum — Patients will chew nicotine gum 3 times a day until discharge or 7 days, whichever comes first
  Other Names: Nicorrete gum
  Arms: Nicotine gum
Other: Regular chewing gum — Patients will chew regular sugar-free gum 3 times a day until discharge or 7 days, whichever comes first
  Other Names: Sugarlees chewing gum
  Arms: regular chewing gum

SUMMARY:
The purpose of this study is to evaluate whether the use of nicotine gum in the postoperative period influences surgical outcome in patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
The main hypothesis of this study is that use of nicotine gum after colorectal surgery will accelerate recovery of bowel function. Eligible patients include all patients undergoing segmental small bowel or large bowel resection with a planned primary anastomosis, planned removal of the nasogastric tube at the end of the surgery, and administration of clear liquids on post-operative day one. Patients who have an ileostomy or colostomy created will be excluded. Patients enrolled in the study will be randomized to one of three groups: nicotine gum, regular gum, or no gum. Patients randomized to nicotine gum or regular gum will chew the gum three times a day for 1 week. The main outcome measure is time to first bowel movement or flatus.

ELIGIBILITY:
Inclusion Criteria:

* Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
* Due to undergo small and/or large partial bowel resection via laparotomy or laparoscopy;

Exclusion Criteria:

* Prior intestinal surgery
* Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures
* American Society of Anesthesiologists (ASA) Class IV or V;
* History of abdominal carcinomatosis;
* History of radiation enteritis;
* Children < 18 or adults > 85 years of age
* Pregnant women
* Current cigarette, cigar smokers and chewers of tobacco. ex smokers who quit less than 3 months ago.
* Patients requiring postoperative ventilation, pressor requirement or ICU stay
* Patients with prior cardiovascular disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ERIC G WEISS, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum
Started | 2 | 2 | 0
Completed | 2 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum | Total
Number analyzed (Participants) | 2 | 2 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 1 | 1 |  | 2
  >=65 years | 1 | 1 |  | 2
Age, Continuous [Mean (Full Range); unit: years] | 58 [48 to 69] | 66 [57 to 76] |  | 62 [48 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  | 1
  Male | 1 | 2 |  | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Bowel Function Recovery
Description: Time to first bowel movement or flatus
Time Frame: 7 days
Measure: Mean (Full Range); unit: days
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum
Number analyzed (Participants) | 2 | 2 | 0
days | 4 [3 to 5] | 5 [4 to 6] |

2. Secondary Outcome: Hospital Stay
Description: Length of postoperative hospital stay
Time Frame: 30 days
Measure: Mean (Full Range); unit: days
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum
Number analyzed (Participants) | 2 | 2 | 0
days | 7 [5 to 9] | 8 [7 to 9] |

3. Secondary Outcome: Post-operative Vomiting
Description: Episodes of vomiting
Time Frame: 30 days
Measure: Mean (Full Range); unit: vomiting episodes
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum
Number analyzed (Participants) | 2 | 2 | 0
vomiting episodes | 0 [0 to 0] | 0 [0 to 0] |

4. Secondary Outcome: Use of NG Tubes
Description: Nasogastric tube (re)insertions
Time Frame: 30 days
Measure: Mean (Full Range); unit: NG Tubes use
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum
Number analyzed (Participants) | 2 | 2 | 0
NG Tubes use | 0 [0 to 0] | 1 [0 to 1] |

ADVERSE EVENTS:
Time Frame: 30 days after procedure
Arm/Group | Nicotine Gum | Regular Chewing Gum | No Gum
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Gum (N=2) | Regular Chewing Gum (N=2) | No Gum (N=0)
Prolonged hospital stay (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Post-operative ileus
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Gum (N=2) | Regular Chewing Gum (N=2) | No Gum (N=0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Low creatinine level (Metabolism and nutrition disorders) | 1 (3) | 1 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglicemia (Metabolism and nutrition disorders) | 1 (5) | 2 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
Principal Investigator decided for an early termination of the enrollment period due to small numbers of subjects consented, with limited data to make conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes